CLINICAL TRIAL: NCT03740113
Title: Kids SipSmartER: A Multi-level Behavioral and Health Literacy Intervention to Reduce Sugar-sweetened Beverages Among Appalachian Middle-school Students
Brief Title: Kids SipSmartER, an Intervention to Reduce Sugar-sweetened Beverages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jamie Zoellner, PhD RD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018019500
Record Dates: First submitted 2018-11-09; First posted 2018-11-14 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Sugary Beverages
Keywords: Sugar sweetened beverages; health disparities; Appalachia

STUDY DESIGN:
Intervention Model Description: Cluster randomized design of schools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kids SipSmartER (Experimental): Kids SIPsmartER is a 12 session, 6-month program with an integrated two-way short service message (SMS) strategy to engage caregivers in SSB role modeling and supporting home SSB environment changes
  Interventions: Behavioral: Kids SipSmartER
- Control (No Intervention): Control arm receives no intervention

INTERVENTIONS:
Behavioral: Kids SipSmartER — Kids SIPsmartER is grounded by the Theory of Planned Behavior as well as health literacy, media literacy, numeracy, and public health literacy concepts
  Arms: Kids SipSmartER

SUMMARY:
Overall Goal: To determine the effectiveness of Kids SIPsmartER in improving sugar-sweetened beverages behaviors among 7th grade students. Secondary aims are to determine (1) changes in secondary student outcomes (e.g. quality of life, BMI z-score, theory-related variables, health and media literacy), (2) changes in caregiver SSB behaviors and home environment, (3) maintenance of outcomes at 19-months post-baseline, (4) assess the reach and representativeness of Kids SIPsmartER, among students and caregivers, and (5) implementation, adoption, and maintenance among teachers and schools.

DETAILED DESCRIPTION:
The intake of sugar-sweetened beverages (SSB, e.g., soda/pop, sweet tea, sports and energy drinks, fruit drinks) is disproportionately high in Appalachia, including among adolescents whose intake is more than double the national average and more than four times the recommended daily amount. There are strong and consistent scientific data and systematic reviews documenting relationships among high SSB consumption and numerous chronic health conditions such obesity, some types of obesity-related cancers, diabetes, cardiovascular disease, and dental erosion and decay. Reaching adolescents with behaviorally-focused health programs where they spend the majority of their time, at school, shows promise. However, engaging caregivers who serve as their child's most influential role model as well as the gatekeeper for the home environment may be equally as important in changing adolescents' SSB behaviors. Finally, there is a great need to understand how to support schools and teachers to deliver and maintain evidence-based health education programs, especially among rural schools. Thus, the overarching goal of this proposal is to work in partnership with Appalachian middle schools to implement and evaluate Kids SIPsmartER. Kids SIPsmartER is a 6-month, school-based, behavior and health literacy curriculum aimed at improving SSB behaviors among middle school students. The program also integrates a two-way short service message (SMS) strategy to engage caregivers in SSB role modeling and supporting home SSB environment changes. Kids SIPsmartER is grounded by the Theory of Planned Behavior as well as health literacy, media literacy, numeracy, and public health literacy concepts. In the proposed cluster-randomized controlled trial, the investigators target 12 middle schools in medically underserved Appalachian counties in southwest Virginia. This study is guided by the RE-AIM (reach, adoption, effectiveness, implementation, and maintenance) framework and is a type 1 hybrid design. The primary aim is to assess changes in SSB behaviors at 7-months among 7th grade students at schools receiving Kids SIPsmartER, as compared to control schools. The investigators will also evaluate changes in secondary student outcomes (e.g., BMI, quality of life, theory-related variables), changes in caregiver outcomes (e.g., SSB behaviors, home SSB environment), and 19-month maintenance of outcomes. The reach and representativeness of Kids SIPsmartER will be assessed. Furthermore, the investigators will use a mixed-methods approach with interviews, surveys, observation, and process evaluation strategies to determine the degree to which teachers implement Kids SIPsmartER as intended and the potential for institutionalization within the schools. The long-term goal of this health promotion and prevention line of research is to establish an effective, scalable, and sustainable multi-level strategy to improve SSB behaviors and reduce SSB-related health inequities and chronic conditions (e.g. obesity, cancer, type II diabetes, heart disease, dental caries) in rural Appalachia.

ELIGIBILITY:
Inclusion Criteria:

* 7th grade students in the 12 enrolled schools during the years their school is randomized to one of these cohorts are eligible to participate
* Parents/caregivers of enrolled middle school students

Exclusion Criteria:

* Data from students with major cognitive disabilities that could compromise self-report behavioral data quality will be excluded

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2024-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirkpatrick BM, Brock DP, Reid AL, Porter KJ, Markwalter TH, You W, Chow PI, Ritterband L, Zoellner J. An SMS intervention to reduce caregiver's sugar-sweetened beverages: impacts on theoretical constructs and parenting practices from a randomized controlled trial in rural appalachia. J Nutr Sci. 2025 Dec 19;14:e91. doi: 10.1017/jns.2025.10057. eCollection 2025. PMID 41496860
- [Derived] Porter KJ, Reid AL, Markwalter T, Kirkpatrick BM, Walters HG, Helms CE, Salyers L, Zoellner JM. Using implementation strategies to promote the maintenance of Kids SIPsmartER in rural Appalachian middle schools: a process evaluation. BMC Public Health. 2025 Jul 3;25(1):2324. doi: 10.1186/s12889-025-23554-x. PMID 40611074
- [Derived] Zoellner JM, Porter KJ, Reid A, Markwalter T, Kirkpatrick B, Brock DP, You W. Comparison of Researcher-Led versus Teacher-Led effectiveness and fidelity: A Hybrid Type 1 study of Kids SIPsmartER in Appalachia middle schools. Transl Behav Med. 2024 Oct 6;14(10):578-587. doi: 10.1093/tbm/ibae041. PMID 39236080
- [Derived] Zoellner JM, You W, Porter K, Kirkpatrick B, Reid A, Brock D, Chow P, Ritterband L. Kids SIPsmartER reduces sugar-sweetened beverages among Appalachian middle-school students and their caregivers: a cluster randomized controlled trial. Int J Behav Nutr Phys Act. 2024 Apr 25;21(1):46. doi: 10.1186/s12966-024-01594-7. PMID 38664715
- [Derived] Yuhas M, Brock DP, Ritterband LM, Chow PI, Porter KJ, Zoellner JM. Retention and engagement of rural caregivers of adolescents in a short message service intervention to reduce sugar-sweetened beverage intake. Digit Health. 2023 Mar 16;9:20552076231160324. doi: 10.1177/20552076231160324. eCollection 2023 Jan-Dec. PMID 36949896
- [Derived] Zoellner JM, Porter KJ, You W, Chow PI, Ritterband LM, Yuhas M, Loyd A, McCormick BA, Brock DP. Kids SIPsmartER, a cluster randomized controlled trial and multi-level intervention to improve sugar-sweetened beverages behaviors among Appalachian middle-school students: Rationale, design & methods. Contemp Clin Trials. 2019 Aug;83:64-80. doi: 10.1016/j.cct.2019.06.011. Epub 2019 Jun 21. PMID 31233859

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Schools
Groups:
- Kids SipSmartER: Kids SIPsmartER is a 12 session, 6-month program with an integrated two-way short service message (SMS) strategy to engage caregivers in sugar-sweetened beverage (SSB) role modeling and supporting home SSB environment changes
  Kids SipSmartER: Kids SIPsmartER is grounded by the Theory of Planned Behavior as well as health literacy, media literacy, numeracy, and public health literacy concepts
Period: Overall Study
Arm/Group | Kids SipSmartER | Control
Started | 547; 6 Schools | 466; 6 Schools
Student Started | 357; 6 Schools | 308; 6 Schools
Caregiver Started | 190; 6 Schools | 158; 6 Schools
Student Completed | 329; 6 Schools | 258; 6 Schools
Caregiver Completed | 126; 6 Schools | 110; 6 Schools
Completed | 455; 6 Schools | 368; 6 Schools
Not Completed | 92; 0 Schools | 98; 0 Schools

BASELINE CHARACTERISTICS:
Population: Analysis population are enrolled students and caregivers who completed the baseline and 7 month assessments
Units Other Than Participants: Schools
Groups:
- Total: Total of all reporting groups
Arm/Group | Kids SipSmartER | Control | Total
Number analyzed (Participants) | 424 | 322 | 746
Number analyzed (Schools) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Total number includes Student and Caregiver participants numbers combined
  years
    Student Age (years): number analyzed (Participants) | 306 | 220 | 526
    Student Age (years) | 12.6 (0.5) | 12.7 (0.4) | 12.7 (0.5)
    Caregiver Age (years): number analyzed (Participants) | 118 | 102 | 220
    Caregiver Age (years) | 40.8 (7.0) | 40.4 (6.2) | 40.6 (6.7)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Total number includes Student and Caregiver participants numbers combined
  Participants
    Student Gender: number analyzed (Participants) | 306 | 220 | 526
    Student Gender: Female | 182 | 107 | 289
    Student Gender: Male | 122 | 109 | 231
    Student Gender: Other or unknown | 2 | 4 | 6
    Caregiver Gender: number analyzed (Participants) | 118 | 102 | 220
    Caregiver Gender: Female | 112 | 96 | 208
    Caregiver Gender: Male | 6 | 6 | 12
    Caregiver Gender: Other or unknown | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total number of participants includes the combination of student and caregiver participants within each arm of the study.
  Participants
    Student Ethnicity: number analyzed (Participants) | 306 | 220 | 526
    Student Ethnicity: Hispanic or Latino | 15 | 9 | 24
    Student Ethnicity: Not Hispanic or Latino | 291 | 211 | 502
    Student Ethnicity: Unknown or Not Reported | 0 | 0 | 0
    Caregiver Ethnicity: number analyzed (Participants) | 118 | 102 | 220
    Caregiver Ethnicity: Hispanic or Latino | 1 | 0 | 1
    Caregiver Ethnicity: Not Hispanic or Latino | 117 | 102 | 219
    Caregiver Ethnicity: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total number includes Student and Caregiver participants numbers combined
  Participants
    Student Race: number analyzed (Participants) | 306 | 220 | 526
    Student Race: American Indian or Alaska Native | 42 | 32 | 74
    Student Race: Asian | 6 | 6 | 12
    Student Race: Native Hawaiian or Other Pacific Islander | 3 | 4 | 7
    Student Race: Black or African American | 9 | 10 | 19
    Student Race: White | 235 | 155 | 390
    Student Race: More than one race | 0 | 0 | 0
    Student Race: Unknown or Not Reported | 11 | 13 | 24
    Caregiver Race: number analyzed (Participants) | 118 | 102 | 220
    Caregiver Race: American Indian or Alaska Native | 1 | 0 | 1
    Caregiver Race: Asian | 2 | 1 | 3
    Caregiver Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Caregiver Race: Black or African American | 3 | 4 | 7
    Caregiver Race: White | 105 | 88 | 193
    Caregiver Race: More than one race | 0 | 0 | 0
    Caregiver Race: Unknown or Not Reported | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 424 | 322 | 746
BMI status [Count of Participants; unit: Participants] — BMI percentile for children is a standardized measure used to assess body weight relative to height, adjusted for age and sex. It is calculated by deriving the Body Mass Index (BMI) from weight (kg) divided by height squared (m²) and then comparing the value to age- and sex-specific growth charts established by the Center for Disease Control.
  Caregiver BMI was calculated from height and weight data using the following equation: kg/m^2 Population: Total number includes Student and Caregiver participants numbers combined
  Participants
    Student BMI Status: number analyzed (Participants) | 306 | 220 | 526
    Student BMI Status: Underweight (student BMI < 5th%; caregiver BMI < 18.5 kg/m2) | 5 | 4 | 9
    Student BMI Status: Healthy Weight (student BMI 5th- <85th%; caregiver BMI 18.5-24.9 kg/m2) | 142 | 103 | 245
    Student BMI Status: Overweight (student BMI 85th-<95th%; caregiver BMI 25-29.9 kg/m2) | 57 | 39 | 96
    Student BMI Status: Obese (student BMI 95th -<99th%; caregiver BMI 30-34.9 kg/m2) | 58 | 40 | 98
    Student BMI Status: Severe Obesity (student BMI >/= 99th%; caregiver BMI >/= 30 kg/m2) | 33 | 15 | 48
    Student BMI Status: Other or unknown | 11 | 19 | 30
    Caregiver BMI Status: number analyzed (Participants) | 118 | 102 | 220
    Caregiver BMI Status: Underweight (student BMI < 5th%; caregiver BMI < 18.5 kg/m2) | 1 | 3 | 4
    Caregiver BMI Status: Healthy Weight (student BMI 5th- <85th%; caregiver BMI 18.5-24.9 kg/m2) | 16 | 28 | 44
    Caregiver BMI Status: Overweight (student BMI 85th-<95th%; caregiver BMI 25-29.9 kg/m2) | 31 | 27 | 58
    Caregiver BMI Status: Obese (student BMI 95th -<99th%; caregiver BMI 30-34.9 kg/m2) | 26 | 16 | 42
    Caregiver BMI Status: Severe Obesity (student BMI >/= 99th%; caregiver BMI >/= 30 kg/m2) | 34 | 21 | 55
    Caregiver BMI Status: Other or unknown | 10 | 7 | 17
Student BMI z-score [Mean (Standard Deviation); unit: z-score] — BMI z-score was calculated using the World Health Organization (WHO) growth reference standards. The z-score represents the number of standard deviations a child's BMI is from the population mean for age and sex. A z-score of 0 corresponds to the median BMI of the reference population. Positive values indicate a BMI higher than the reference median, while negative values indicate a BMI lower than the reference median. Higher z-scores generally indicate increased adiposity, with standard clinical thresholds defining overweight as a BMI z-score ≥ 1 and obesity as a BMI z-score ≥ 2. Population: BMIz-scores are only calculated for the student sample. A total of 11 KSS student participants and 19 control student participants were not weighed and therefore are not in the sample.
  z-score
    number analyzed (Participants) | 295 | 201 | 496
    (all) | 0.9 (1.1) | 1.0 (1.0) | 0.9 (1.1)
Student BMI percentile [Mean (Standard Deviation); unit: percentile] — BMI percentile for children is a standardized measure used to assess body weight relative to height, adjusted for age and sex. It is calculated by deriving the Body Mass Index (BMI) from weight (kg) divided by height squared (m²) and then comparing the value to age- and sex-specific growth charts established by the CDC. Population: BMI percentiles are only calculated for the student sample. A total of 11 KSS student participants and 19 control student participants were not weighed and therefore are not in the sample.
  percentile
    number analyzed (Participants) | 295 | 201 | 496
    (all) | 73.2 (27.1) | 75.8 (24.6) | 74.1 (26.2)
Caregiver Educational Attainment [Count of Participants; unit: Participants] — Population: Only caregivers are asked for their educational attainment.
  Participants
    number analyzed (Participants) | 118 | 102 | 220
    High School, GED, or less | 28 | 28 | 56
    Some college, Associates degree | 49 | 36 | 85
    4-year college degree or higher | 36 | 35 | 71
    Other or unknown | 5 | 3 | 8
Caregiver Household Income [Count of Participants; unit: Participants] — Population: Only caregivers are asked to report their family's annual household income
  Participants
    number analyzed (Participants) | 118 | 102 | 220
    <$25,000 | 20 | 18 | 38
    $25,000-$49,000 | 16 | 20 | 36
    $50,000-$74,999 | 25 | 18 | 43
    >/= $75,000 | 37 | 31 | 68
    Other or unknown | 20 | 15 | 35
Caregiver BMI [Mean (Standard Deviation); unit: kg/m2] — Population: Only caregivers weight and height were calculated into a BMI. Additionally, a total of 10 KSS caregiver participants and 7 caregiver control participants did not report their weights and heights so BMI could not be calculated for them.
  kg/m2
    number analyzed (Participants) | 108 | 95 | 203
    (all) | 32.1 (7.7) | 29.5 (8.0) | 30.8 (7.9)

OUTCOME MEASURES:

1. Primary Outcome: Student: SSB Change From Baseline to 7-months (All Participants)
Description: Change in ounces of sugar sweetened beverage consumption from Baseline to 7-months as measured via the validated Beverage Intake Questionnaire (BEVQ-15). Participants were asked to report how often and how much of the following sugary drinks they consumed in the past 30 days: regular soft drinks, sweetened juice beverage/drink, sweetened tea, coffee with sugar, energy/sports drinks. Using standardized and validated scoring procedures, daily totals for each of the sugary beverages were determined by multiplying intake frequency by portion size. These daily total intakes were then summed across the five sugary drink types to obtain a total daily intake, in fluid ounces, of all sugary drinks. Change scores were calculated by subtracting the baseline sugary drink intake from the 7 month follow-up.
Time Frame: Baseline and 7-months
Population: This analysis only includes student participants. While caregivers were analyzed for change in SSB, caregiver SSB change was a secondary outcome and therefore they are not reported here. Overall participants analyzed includes students who completed both the baseline and 7 month follow up items for the BEVQ-15.
Measure: Mean (95% Confidence Interval); unit: fluid ounces
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 306 | 220
fluid ounces | -9.9 [-12.2 to -7.6] | -2.7 [-5.4 to -0.1]

2. Secondary Outcome: Caregiver: SSB Change From Baseline to 7-months (All Participants)
Description: as for outcome 1
Time Frame: Baseline and 7-months
Population: This analysis only includes caregiver participants. While students were analyzed for change in SSB, student SSB change was a primary outcome and therefore they are not reported here. Overall participants analyzed includes caregivers who completed both the baseline and 7 month follow up items for the BEVQ-15.
Measure: Mean (80% Confidence Interval); unit: fluid ounces
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 118 | 102
fluid ounces | -8.2 [-12.3 to -4.1] | -6.3 [-11.3 to -1.3]

3. Secondary Outcome: Student: BMI Z-score Change From Baseline to 7-months
Description: Student BMI z-score: BMI z-score was calculated using the World Health Organization (WHO) growth reference standards. The z-score represents the number of standard deviations a child's BMI is from the population mean for age and sex. A z-score of 0 corresponds to the median BMI of the reference population. Positive values indicate a BMI higher than the reference median, while negative values indicate a BMI lower than the reference median. Higher z-scores generally indicate increased adiposity, with standard clinical thresholds defining overweight as a BMI z-score ≥ 1 and obesity as a BMI z-score ≥ 2.
Time Frame: Baseline and 7-months
Population: Because BMI is calculated differently for adults, this analysis only includes student participants. Caregiver BMI changes are reported separately. Overall participants analyzed includes students who completed both the baseline and 7 month height and weight measures.
Measure: Mean (95% Confidence Interval); unit: z-score
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 295 | 166
z-score | 0.02 [-0.01 to 0.05] | -0.018 [-0.09 to 0.06]

4. Secondary Outcome: Caregiver: BMI Change From Baseline to 7-Months
Description: Caregiver BMI was calculated from height and weight data using the following equation: kg/m^2
Time Frame: Baseline and 7-months
Population: Because BMI is calculated differently for children, this analysis only includes caregiver participants. Student BMI changes are reported separately. Overall participants analyzed includes caregivers who reported their baseline and 7 month height and weight measures.
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 105 | 92
kg/m^2 | -0.3 [-0.6 to -0.1] | -0.65 [-1.0 to -0.3]

5. Secondary Outcome: Student and Caregiver: Quality of Life Change From Baseline to 7-months--Overall Health Rating
Description: Overall health rating is a Single item question asking to rate general overall health and scored on a 5-point Likert scale from 1=poor to 5=excellent.
Time Frame: Baseline and 7-months
Population: Overall participants analyzed includes students and caregivers who completed both the baseline and 7 month overall health rating item.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 422 | 311
units on a scale
  Students: Overall Health Rating Change: number analyzed (Participants) | 307 | 214
  Students: Overall Health Rating Change | 0.06 [0.003 to 0.1] | 0.03 [-0.1 to 0.2]
  Caregivers: Overall Health Rating Change: number analyzed (Participants) | 115 | 97
  Caregivers: Overall Health Rating Change | 0.04 [-0.0 to 0.1] | -0.06 [-0.2 to 0.1]

6. Secondary Outcome: Caregiver: Quality of Life Change From Baseline to 7-months--Unhealthy Days
Description: Using validated scoring procedures, an unhealthy days score was computed by adding the number of physically and mentally unhealthy days within the past 30 days, with a minimum score of 0 and maximum score of 30 days. Higher scores indicate worse quality of life.
Time Frame: Baseline and 7-months
Population: Questions were only asked of caregiver and students are not included in the analysis. Overall participants analyzed includes caregivers who completed both the baseline and 7-month follow up items for the quality of life scale.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 109 | 93
units on a scale | -0.3 [-1.1 to 0.6] | -1.7 [-4.3 to 0.9]

7. Secondary Outcome: Student: Quality of Life Change From Baseline to 7-months--school Related Function
Description: School-related quality of life (QOL) was assessed with the 5-item school functioning subscale of the Pediatric QOL Inventory which used a 5-point Likert scale (i.e., 1 = never a problem, 5 = almost always a problem). Applying validated scoring procedures, items were reverse-scored and linearly transformed to a 0 to 100 scale with higher scores indicating higher school-related QOL.
Time Frame: Baseline and 7-months
Population: This analysis only includes student participants. Caregiver quality of life measures are reported separately. Overall participants analyzed includes students who completed both the baseline and 7 month school related function items.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 294 | 211
units on a scale | -1.7 [-3.9 to 0.4] | -3.9 [-7.0 to -.07]

8. Post Hoc Outcome: Caregiver: SSB Change From Baseline to 7-months for Caregivers Consuming > 24 fl oz SSB at Baseline
Description: as for outcome 1
Time Frame: Baseline and 7-months
Population: This analysis only includes caregiver participants who consumed > 24 fluid ounces of SSB at Baseline AND who completed both the Baseline and 7 month SSB items for the BEVQ-15. While students were analyzed similarly, student SSB change across Baseline SSB intake was a primary outcome and therefore they are not reported here.
Measure: Mean (95% Confidence Interval); unit: fluid ounces
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 33 | 28
fluid ounces | -23.7 [-29.7 to -17.7] | -9.8 [-13.6 to -6.1]

9. Post Hoc Outcome: Caregiver: SSB Change From Baseline to 7-months for Caregivers Consuming > 12 fl oz SSB at Baseline
Description: as for outcome 1
Time Frame: Baseline and 7-months
Population: This analysis only includes caregiver participants who consumed > 12 fluid ounces of SSB at Baseline AND who completed both the Baseline and 7 month SSB items for the BEVQ-15. While students were analyzed similarly, student SSB change across Baseline SSB intake was a primary outcome and therefore they are not reported here.
Measure: Mean (95% Confidence Interval); unit: fluid ounces
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 58 | 50
fluid ounces | -17.5 [-20.8 to -14.2] | -7.1 [-9.1 to -5.1]

10. Post Hoc Outcome: Caregiver: SSB Change From Baseline to 7-months for Caregivers Consuming > 8 fl oz SSB at Baseline
Description: as for outcome 1
Time Frame: Baseline and 7-months
Population: This analysis only includes caregiver participants who consumed > 8 fluid ounces of SSB at Baseline AND who completed both the Baseline and 7 month SSB items for the BEVQ-15. While students were analyzed similarly, student SSB change across Baseline SSB intake was a primary outcome and therefore they are not reported here.
Measure: Mean (95% Confidence Interval); unit: fluid ounces
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 70 | 58
fluid ounces | -15.0 [-18.6 to -11.5] | -5.8 [-7.2 to -4.5]

11. Post Hoc Outcome: Student: SSB Change From Baseline to 7-months for Students Consuming > 24 fl oz SSB at Baseline
Description: as for outcome 1
Time Frame: Baseline and 7-months
Population: This analysis only includes student participants who consumed > 24 fluid ounces of SSB at Baseline AND who completed both the Baseline and 7 month SSB items for the BEVQ-15. While caregivers were analyzed similarly, caregiver SSB change across Baseline SSB intake was a secondary outcome and therefore they are not reported here.
Measure: Mean (95% Confidence Interval); unit: fluid ounces
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 141 | 82
fluid ounces | -23.0 [-27.0 to -19.0] | -10.3 [-17.7 to -2.9]

12. Post Hoc Outcome: Student: SSB Change From Baseline to 7-months for Students Consuming > 12 fl oz SSB at Baseline
Description: as for outcome 1
Time Frame: Baseline and 7-months
Population: This analysis only includes student participants who consumed > 12 fluid ounces of SSB at Baseline AND who completed both the Baseline and 7 month SSB items for the BEVQ-15. While caregivers were analyzed similarly, caregiver SSB change across Baseline SSB intake was a secondary outcome and therefore they are not reported here.
Measure: Mean (95% Confidence Interval); unit: fluid ounces
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 213 | 136
fluid ounces | -15.5 [-19.0 to -12.0] | -7.4 [-11.2 to -3.7]

13. Post Hoc Outcome: Student: SSB Change From Baseline to 7-months for Students Consuming > 8 fl oz SSB at Baseline
Description: as for outcome 1
Time Frame: Baseline and 7-months
Population: This analysis only includes student participants who consumed > 8 fluid ounces of SSB at Baseline AND who completed both the Baseline and 7 month SSB items for the BEVQ-15. While caregivers were analyzed similarly, caregiver SSB change across Baseline SSB intake was a secondary outcome and therefore they are not reported here.
Measure: Mean (95% Confidence Interval); unit: fluid ounces
Arm/Group | Kids SipSmartER | Control
Number analyzed (Participants) | 247 | 160
fluid ounces | -13.5 [-16.2 to -10.8] | -5.7 [-8.5 to -2.9]

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the 19-month follow-up data collection
Description: Given the low risk nature of the sugary beverage intervention, adverse event and/or serious adverse event were determined in non-systematic method, including self-reporting by participants.
Arm/Group | Kids SipSmartER | Control
All-Cause Mortality (participants affected / at risk) | 0/424 | 0/322
Serious Adverse Events (participants affected / at risk) | 0/424 | 0/322
Other Adverse Events (participants affected / at risk) | 0/424 | 0/322

LIMITATIONS AND CAVEATS:
1. The unique rural Appalachian sample may limit generalizability
2. Uncontrollable study disruptions caused by COVID-19 required different survey data collection protocols at some schools and halted enrollment of new schools in the 2020-2021
3. COVID-19 related impacts related to lower study retention (Spring 2020) and enrollment (2021-2022)
4. Caregivers' self-reported weight
5. Research staff were not blinded to schools' randomized allocation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT03740113/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT03740113/SAP_001.pdf